CLINICAL TRIAL: NCT00351117
Title: A Randomized, Placebo-controlled Trial of St.John's Wort(a Natural Health Product) in the Treatment on Raynaud's Phenomenon
Brief Title: St. John's Wort in the Treatment of Raynaud's Phenomenon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Janet Pope, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-06-355; 250347647
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Raynaud's Disease
Keywords: St. John's Wort; Selective Serotonin Receptor Inhibitor; Microvasculature; Natural Health Products
MeSH Terms: conditions — Raynaud Disease | interventions — Hypericum extract LI 160; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): St. John's wort 300mg PO TID
  Interventions: Drug: St. John's Wort
- 2 (Placebo Comparator): Lactose in capsule matching the St. John's wort. 300mg PO TID
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: St. John's Wort — SJW in capsule form 300 mg PO TID
  Other Names: Webber natural brand, product number 5006.
  Arms: 1
Drug: Lactose — lactose in gelatin capsule that same as St. John's wort
  Arms: 2

SUMMARY:
This trial will test the efficacy of St. John's Wort (SJW) as a supplement, in the treatment of Raynaud's phenomenon (RP). The investigators are hypothesizing that taking SJW 300mg, 3 times a day will decrease the frequency, duration, and severity of RP attacks when compared to placebo.

Patients with RP will answer questionnaires and self-evaluate their symptoms of RP as a baseline. Then they will be assigned to either a treatment (will receive SJW capsules) or placebo (will receive non-therapeutic capsules) group. They will be required to take their capsules, self-evaluate their progress and be evaluated every two weeks in a clinic. The treatment phase will last six weeks.

This trial will be conducted in a way to mimic the normal usage of natural products. Patients will not be required to stop any current treatment for RP.

DETAILED DESCRIPTION:
Raynaud's Phenomenon (RP) is a common vasospastic problem of digital artery vessels causing pain and ischemic fingers (the fingers turn white and then blue and or red). It is considered primary when it is not associated with other conditions. Raynaud's symptoms that are associated with pathological underlying cause especially connective tissue diseases are defined as secondary Raynaud's and are usually more severe than primary symptoms. Selective Serotonin receptor inhibitors (SSRIs) have shown to be effective in decreasing the symptoms of RP.

St. John's Wort (SJW) is an natural product that is presently approved by Health Canada for treatment of depression. It is believed that SJW would have mechanism of action very similar to SSRIs.

This clinical trial will measure the efficiency of SJW in decreasing the frequency, duration and severity of RP attacks. SJW will be test as a supplement to other treatments already in place. 76 patients (38 with primary Raynaud's and half with secondary Raynaud's) will be recruited from the Rheumatology clinic of St. Joseph's Health Care in London, Ontario. The recruitment period will span 18 months. As they enter the trial, subjects will be assigned to a treatment or a placebo group according to a pre-set randomization schedule. This assignment will be stratified for primary or secondary Raynaud's and double-blinded (patient and investigator).

The primary outcome measure (frequency, duration and severity) will be assessed by the patient on a daily basis using a journal provided by the investigator. Secondary outcome measures will include functions questionnaires (HAQ, SF-36, DASH) and biological markers of endothelial damage (V-CAM, I-CAM, VEGF, von Willebrand factor), will be conducted as a baseline and at the conclusion of the treatment phase.

Patients participation will span 8-10 weeks. The first two weeks are a baseline measurement for the status of RP using the journals, questionnaires, and serum tests. The treatment period will last 6 weeks in which the subject will be taking the capsules that they have been assigned and will be evaluated for changes or side-effects every two weeks. At the last visit the questionnaires and serum test will be repeated.

Other results which may arise from the trial are:

* The safety of SJW in rheumatology patients, by monitoring side-effects
* The attitude of rheumatology patients in using Natural Health Products, by a questionnaire
* Elucidating parts of the RP mechanism, by measuring bio-markers
* Differences between primary and secondary RP, by stratified randomization

The results will be analyzed for all three primary outcome measures as a difference of between baseline and treatment. These differences will be compared between treatment and placebo and each will be stratified for primary vs. secondary and possibly other demographic data.

This trial, if positive, will offer another treatment to RP patients. This option will possibly have less side-effects and be better accepted because it is a Natural Product.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females between 16 and 70 years old
* Primary or secondary Raynaud's phenomenon, as diagnosed by a rheumatologist
* Clinical need for treatment of Raynaud's phenomenon
* Experiences at least 7 attacks per week
* Willing and able to provide informed consent

Exclusion Criteria:

* Prior allergic reaction to St. John's Wort
* Pregnancy or possibility or pregnancy in the next 4 months
* Women that are currently breastfeeding
* Depression requiring treatment
* Use of SSRIs or other antidepressants with the exception of low dose amitriptyline used for reasons other than depression
* Use of drugs that are potentiated by St. John's Wort, such as cyclosporine, coumadin, digoxin, and theophylline. The complete list of contraindicated medications can be received from investigator
* Clinically significant non-compliance with past therapies
* Anticipated need for surgery (sympathectomy) in the next three months

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Frequency of Raynaud's Phenomenon (RP) attacks | 6 weeks
Duration of RP attacks | 6 weeks
Severity of RP attacks | 6 weeks

SECONDARY OUTCOMES:
Daily functions questionnaires (HAQ, SF-36, DASH) | 6 weeks
Biological markers of endothelial damage (V-CAM, I-CAM, VEGF, etc.) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD, MPH, Principal Investigator — Associate Professor of Medicine University of Western Ontario
Locations (1):
- Rheumatology Clinic, St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Background] Schrader E. Equivalence of St John's wort extract (Ze 117) and fluoxetine: a randomized, controlled study in mild-moderate depression. Int Clin Psychopharmacol. 2000 Mar;15(2):61-8. doi: 10.1097/00004850-200015020-00001. PMID 10759336
- [Background] Coleiro B, Marshall SE, Denton CP, Howell K, Blann A, Welsh KI, Black CM. Treatment of Raynaud's phenomenon with the selective serotonin reuptake inhibitor fluoxetine. Rheumatology (Oxford). 2001 Sep;40(9):1038-43. doi: 10.1093/rheumatology/40.9.1038. PMID 11561116
- [Background] Pope J. Raynaud's phenomenon (primary). Clin Evid. 2003 Jun;(9):1339-48. No abstract available. PMID 12967424
- [Background] Bolte MA, Avery D. Case of fluoxetine-induced remission of Raynaud's phenomenon--a case report. Angiology. 1993 Feb;44(2):161-3. doi: 10.1177/000331979304400213. No abstract available. PMID 8434812
- [Background] Brenner R, Azbel V, Madhusoodanan S, Pawlowska M. Comparison of an extract of hypericum (LI 160) and sertraline in the treatment of depression: a double-blind, randomized pilot study. Clin Ther. 2000 Apr;22(4):411-9. doi: 10.1016/S0149-2918(00)89010-4. PMID 10823363
- [Background] Pope JE, Prashker M, Anderson J. The efficacy and cost effectiveness of N of 1 studies with diclofenac compared to standard treatment with nonsteroidal antiinflammatory drugs in osteoarthritis. J Rheumatol. 2004 Jan;31(1):140-9. PMID 14705233
- [Background] Jaffe IA. Serotonin reuptake inhibitors in Raynaud's phenomenon. Lancet. 1995 May 27;345(8961):1378. doi: 10.1016/s0140-6736(95)92582-1. No abstract available. PMID 7752794
- [Background] Knuppel L, Linde K. Adverse effects of St. John's Wort: a systematic review. J Clin Psychiatry. 2004 Nov;65(11):1470-9. doi: 10.4088/jcp.v65n1105. PMID 15554758
- [Background] Lecrubier Y, Clerc G, Didi R, Kieser M. Efficacy of St. John's wort extract WS 5570 in major depression: a double-blind, placebo-controlled trial. Am J Psychiatry. 2002 Aug;159(8):1361-6. doi: 10.1176/appi.ajp.159.8.1361. PMID 12153829
- See also: American website of institute of arthritis: general medical information on Raynaud's Disease — http://www.NIAMS.NIH.gov/Health_Info/Raynauds_Phenomenon/default.asp
- See also: Canadian complementary and alternative medicine research group: contains details on how to conduct a natural product trials and has a lot of resources. — http://incamresearch.ca
- See also: A database that is linked to MedLine and does searches for herbal medicine only. — http://www.herbmed.org
- See also: Health Canada Natural Health product site: information on regulation and legislature — http://www.hc-sc.gc.ca/dhp-mps/prodnatur/index_e.html